CLINICAL TRIAL: NCT07285603
Title: A Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of M6229 Administered as a 120-hour Continuous Infusion at Three Sequential Dose Levels Versus Placebo in Healthy Subjects
Brief Title: A Study in Healthy Subjects to Assess the Safety and Tolerability of a 120-hour Continuous Infusion of M6229
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Matisse Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: M6229-C002
Record Dates: First submitted 2025-09-29; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects
Keywords: M6229; Unfractioned Heparin; Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M6229 (Experimental): A low-anticoagulant heparin in low, mid, and high dose. IV administration.
  Interventions: Drug: M6229
- Placebo (Placebo Comparator): Saline solution; IV administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M6229 — Continuous 120-hour intravenous infusion of M6229
  Arms: M6229
Drug: Placebo — Continuous 120-hour intravenous infusion of placebo (saline)
  Arms: Placebo

SUMMARY:
This is a Phase I, single-center, randomized, single-blind, placebo-controlled study in healthy subjects assessing the safety, tolerability and pharmacokinetic profile of three different dose levels of M6229 when administered continuously for 120 hours.

DETAILED DESCRIPTION:
Three dose levels of M6229 will be assessed in sequential study cohorts. Each cohort will consist of up to 3 male and 3 female subjects (2 male and 2 female subjects on M6229, 1 male and 1 female subject on placebo). Following a screening period of up to 28 days during which eligibility will be assessed, subjects will be randomized to M6229 or placebo and start a 120-hour continuous infusion on Day 1. Subjects will undergo safety assessments (incl. laboratory assessments) and pharmacokinetic sampling following a predefined schedule from Day 1 until Day 9. Subjects will be discharged on Day 9. The clinical study will be completed with an end-of-study visit, which will take place between 5 to 9 days after the last treatment-defined assessment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male or female, aged 18 - 55 years at time of informed consent
* BMI between 18.0 - 30.0 kg/m2
* Normal vital signs (resting pulse rate and resting blood pressure)
* Normal ECG parameters (PR, QRS, QTc)
* Normal coagulation parameters (aPTT, PTT/INR and thrombin time)
* Female subjects must have a negative serum pregnancy test
* Willing and able to adhere to contraceptive requirements

Exclusion Criteria:

* History of clinically significant medical illness
* Laboratory abnormalities
* Major surgery or trauma in previous 6 months
* Positive test for HIV, HBsAg, or HCV
* History of heart arrhythmias, tachycardia at rest, or history of risk factors for Torsade de Pointes syndrome
* Clinically relevant allergy or drug hypersensitivity (incl. heparin)
* Smokes daily more than 5 cigarettes or equivalent
* History of postural disorders
* Lack of adequate venous access
* Current or ongoing history of urinary retention
* Use of prescription or nonprescription medication within 7 days prior to Day 1
* Received an investigational drug or medical device recently, or >3 investigational agents in last 12 months, or currently enrolled in an investigational study
* Donated blood or substantial blood loss within 60 days prior to Day 1
* Any condition, preplanned surgery or procedure that would interfere with the study conduct and/or with the subject's best interest
* Subject is vulnerable
* Subject is an employee of the investigator, clinical site, or Sponsor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence and type of Adverse Events (AEs) | Until End of Study (Day 14-18)
  Any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Change in electrocardiograms (ECGs) from baseline | Until End of Study (Day 14-18)
  Clinically significant changes in PR interval, QRS interval, QT interval, and QTcF
Change in vital signs - blood pressure | Until End of Study (Day 14-18)
  Changes in systolic and diastolic blood pressure in mmHg
Change in vital signs - pulse rate | Until End of Study (Day 14-18)
  Change in pulse rate measured in beat per minute
Change in vital signs - respiratory rate | Until End of Study (Day 14-18)
  Change in respiratory rate measured in breaths per minute
Change in vital signs - body temperature | Until End of Study (Day 14-18)
  Changes in body temperature measured in degrees Celcius
Pharmacokinetics: Maximum observed analyte concentration (Cmax) | Until Day 9 (192 hours)
Pharmacokinetics: Maximum observed analyte concentration (tmax) | Until Day 9 (192 hours)
Pharmacokinetics: Last measured quantifiable concentration (tlast) | Until Day 9 (192 hours)
Pharmacokinetics: Area under the curve (AUC) | Until Day 9 (192 hours)
Pharmacokinetics: Elimination half-life (t1/2) | Until Day 9 (192 hours)
Pharmacokinetics: Volume of distribution (Vd) | Until Day 9 (192 hours)
Pharmacokinetics: Clearance (Cl) | Until Day 9 (192 hours)
Pharmacokinetics: Amount excreted (Ae) in urine | Until Day 9 (192 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iten PX, Meier M. Beta-hydroxybutyric acid--an indicator for an alcoholic ketoacidosis as cause of death in deceased alcohol abusers. J Forensic Sci. 2000 May;45(3):624-32. PMID 10855969
- [Background] Zimmer KP, Lentze MJ, Nutzenadel W, Rodeck B. On the situation of pediatric gastroenterology in a so-called developed country. J Pediatr Gastroenterol Nutr. 2002 Sep;35(3):241-2. doi: 10.1097/00005176-200209000-00001. No abstract available. PMID 12360993
- See also: Related Info — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2024-512022-28-01